CLINICAL TRIAL: NCT02564692
Title: Alzheimer's Prevention Registry GeneMatch Program
Brief Title: GeneMatch: A Program of the Alzheimer's Prevention Registry to Match Individuals to Studies Based on Apolipoprotein E (APOE) Genotype
Status: Enrolling by invitation | Type: Observational
Sponsor: Banner Health (Other)
Responsible Party: Principal Investigator, Jessica Langbaum, PhD, Senior Director, Research Strategy, Banner Health
Other Study IDs: APR-001
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Alzheimer's Prevention Registry GeneMatch program is to identify a large group of people interested in participating in research studies or clinical trials based in part on their genetic background. This genetic information will be used to match interested individuals to studies, providing a recruitment resource to the Alzheimer's scientific community. Interested individuals should visit www.endALZnow.org/GeneMatch to join the GeneMatch program.

DETAILED DESCRIPTION:
The primary objectives of the Alzheimer's Prevention Registry GeneMatch program are to (1) identify and characterize a large cohort of people who are interested in, and may be eligible to participate in, current and future preclinical Alzheimer's disease research studies and clinical trials based on their genetic background, and (2) provide information to these individuals about research studies for which they may be eligible, based in part on their genetic background. Cognitively unimpaired individuals age 50 to 90, inclusive, are eligible to enroll in GeneMatch. GeneMatch will provide participants with a genetic sample kit (a cheek swab) to test for a specific gene called apolipoproteins E (APOE). GeneMatch does not disclose the results of the APOE test to participants. GeneMatch may use the APOE test results to match participants to research studies. Participants are under no obligation to pursue these study opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-90, inclusive
* Provide basic demographic, medical history, and contact information
* Consent to APOE genotyping without receiving results
* Live in the United States

Exclusion Criteria:

* Unable to comply with this project's protocol requirements
* Self-reported diagnosis of dementia or any other objective cognitive impairment syndrome

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This large research study will ultimately enroll 500,000 adults. We will recruit subjects from all over the United States, as everything is done via email, mail, or/and phone.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2015-11; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of individuals who enroll in GeneMatch | 15 years

SECONDARY OUTCOMES:
Number of individuals referred to research studies | 15 years
Number of individuals who enroll in research studies | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Jessica B Langbaum, PhD, Principal Investigator — Banner Alzheimer's Institute
Locations (1):
- Banner Alzheimer's Institute, Phoenix, Arizona, United States

REFERENCES:
- [Result] Langbaum JB, Karlawish J, Roberts JS, Wood EM, Bradbury A, High N, Walsh TL, Gordon D, Aggarwal R, Davis P, Stowell C, Trisko L, Langlois CM, Reiman EM, Tariot PN. GeneMatch: A novel recruitment registry using at-home APOE genotyping to enhance referrals to Alzheimer's prevention studies. Alzheimers Dement. 2019 Apr;15(4):515-524. doi: 10.1016/j.jalz.2018.12.007. Epub 2019 Feb 13. PMID 30772251